CLINICAL TRIAL: NCT05548192
Title: Evaluation of the SmartPICC System for PICC Placement in Adults: A Safety and Technical Feasibility Study
Brief Title: SmartPICC-1 Feasibility Study Technical Feasibility Study
Status: Completed | Type: Observational
Sponsor: Piccolo Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD-15-325
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Catheter Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: SmartPICC-1 System — The SmartPICC system is indicated for use as an alternative method to chest x-ray or fluoroscopy confirmation of PICC tip placement in adult patients when proper ECG detection is available. The SmartPICC system provides a supplemental intravascular ionic dilution feature that provides qualitative blood flow information to the user to aid catheter navigation during PICC placement.

SUMMARY:
The primary objective of this study is to evaluate the safety and technical feasibility of the Piccolo Medical SmartPICC System, indicated for guidance and positioning of commercially available central venous catheters, for PICC placement in adults.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and technical feasibility of the Piccolo Medical SmartPICC System for PICC placement in adults. The SmartPICC system is indicated for guidance and positioning of commercially available central venous catheters. In this prospective, single arm (non-randomized), safety and technical feasibility study, adult volunteers who meet the protocol entry criteria and are scheduled to undergo PICC placement will be recruited. Immediately following placement with use of the SmartPICC System, subjects will undergo an assessment of the PICC placement site, as technical feasibility will be evaluated as the ability of the SmartPICC System to provide venous navigation for PICC placement in the lower superior vena cava (L-SVC), cavoatrial junction (CAJ), or proximal right atrium (RA) as confirmed by radiologic review. Safety will be evaluated as freedom from serious adverse events (SAEs) directly attributable to the SmartPICC system. Subjects will be evaluated at 12-24 hours post-placement to ensure safety, in addition to a review of subject medical records 7 days post PICC placement.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent, including authorization to release health information
* Subject between 22-85 years of age at the time of consent
* Subject is scheduled for PICC placement
* Subject understands and is able and willing to comply with the study requirements
* Subject has provided a negative pregnancy test (if subject is a woman of childbearing potential (WOCBP))

Exclusion Criteria:

* Contraindicated for PICC
* Subject is enrolled in another clinical study where the safety profile is not yet established or may otherwise confound the SmartPICC-1 Study results
* Subject is deemed ineligible for the study in the opinion of the investigator, physician, and/or PICC nurse
* Subject has single ventricle anatomy
* Subject has a BMI that, in the opinion of the investigator, physician, and/or PICC nurse, would interfere with successful PICC placement
* Subjects with known stenosis of the upper arm and right-side veins that may prevent successful PICC placement
* Subject has mechanical circulatory support device (e.g. ECMO, VAD)
* Subject is pregnant
* Subject has or is suspected to have COVID-19

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects who have been prescribed a PICC
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
SmartPICC placement efficacy | Immediately post procedure
  Technical feasibility will be evaluated as the ability of a SmartPICC System to provide venous navigation for PICC placement in the lower superior vena cava (L-SVC), cavoatrial junction (CAJ), or proximal right atrium (RA) as confirmed by radiologic review.
SmartPICC safety | up to 7 days post procedure
  Safety will be evaluated as freedom from serious adverse events (SAEs) directly attributable to the SmartPICC System. subjects will be evaluated at 12-24 hours post-placement to ensure that no investigational device or investigational procedure related Adverse Events have occurred. A review of subject medical records will also be performed at 7 days post PICC placement to ensure that there was no post procedure phlebitis, thrombosis, or central line-associated bloodstream infection (CLABSI) attributable to the study device.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - El Camino Health - Mountain View, San Francisco, California
  - CPMC Van Ness, San Francisco, California

IPD SHARING:
Plan to Share IPD: Undecided